CLINICAL TRIAL: NCT01184846
Title: A Single-arm Study to Demonstrate the Efficacy and Safety of Privigen in the Treatment of Subjects With Chronic Inflammatory Demyelinating Polyneuropathy (CIDP)
Brief Title: Study of Efficacy and Safety of Privigen in Subjects With Chronic Inflammatory Demyelinating Polyneuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IgPro10_3001; 1504 (Other: CSL Behring); 2009-017672-24 (EudraCT Number)
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Chronic inflammatory demyelinating polyneuropathy; CIDP
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IgPro10 (Experimental): 10% liquid formulation of human immunoglobulin (IgPro10). IgPro10 will be administered by IV infusion as one induction dose of 2 g/kg body weight (bw), followed by seven 3-weekly maintenance doses of 1 g/kg bw.
  Interventions: Biological: 10% liquid formulation of human immunoglobulin

INTERVENTIONS:
Biological: 10% liquid formulation of human immunoglobulin
  Other Names: IgPro10; Privigen

SUMMARY:
The objective of this study is to demonstrate the efficacy and safety of Privigen in subjects with CIDP.

ELIGIBILITY:
Inclusion Criteria:

IVIG-untreated subjects:

* Either subjects with newly diagnosed CIDP (developing over at least 2 months) or subjects with an IVIG treatment interruption for at least 1 year with a progressive disease (deteriorating in the last 2 months) prior to enrolment.
* Actual diagnosis (including electrophysiology) of CIDP with progressive or relapsing dysfunction from motor and sensory or symmetric motor nerve only in at least 1 limb resulting from neuropathy. Criteria for definite or probable CIDP according to EFNS/PNS guideline.
* Age ≥18 years.
* Male or female.
* Written informed consent for study participation obtained before undergoing any study specific procedures.

IVIG-pretreated subjects:

* Being treated regularly with IVIG on a fixed cycle length of 2 to 6 weeks ± 5 days in the last 6 months, on a fixed dosage of ± 20 % in the last 6 months and deteriorating by at least 1 INCAT score point during the Washout Period of up to 10 weeks (except for an increase from 0 to 1 solely due to upper limb score).
* Historic diagnosis of CIDP with progressive or relapsing dysfunction from motor and sensory or symmetric motor nerve only in at least 1 limb resulting from neuropathy. Criteria for definite or probable CIDP according to EFNS/PNS guideline.
* Age ≥18 years.
* Male or female.
* Written informed consent for study participation obtained before undergoing any study specific procedures.

Exclusion Criteria:

* A motor syndrome that fulfils criteria for multifocal motor neuropathy (MMN) with conduction block (i.e., upper limb motor weakness without sensory deficit and with a 50% decrease in action potential amplitude or area on proximal compared with distal stimulation in motor nerves).
* CIDP with monoclonal gammopathy of uncertain significance (CIDP-MGUS) with anti-MGUS antibodies and patients with distal acquired demyelinating symmetric (DADS)neuropathy.
* Any disease (mainly neurological or chronic orthopedic) that may cause symptoms or may interfere with treatment or outcome assessments with the INCAT (e.g., diphtheria, drug or toxin exposure and diabetes mellitus likely to have caused the neuropathy, IgM paraproteinemia, familial neuropathy, borreliosis with radiculopathy, post-polio-syndrome,M. Parkinson, stroke).
* Current malignancy.
* History of cardiac insufficiency (New York Heart Association [NYHA] III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease, congestive heart failure or severe hypertension.
* History of thrombotic episodes (deep vein thrombosis, myocardial infarction, cerebrovascular accident).
* Migraine associated with IVIG infusion in the last 3 months prior to enrolment.
* Known allergic or other severe reactions to blood products including intolerability to previous IVIG (i.e. severe headache, hypersensitivity, intravascular hemolysis).
* Subjects with serum IgA level less than 50% of the lower normal limit.
* Known hyperprolinemia.
* Any condition (including alcohol, drug or medication abuse) that is likely to interfere with evaluation of the study product or satisfactory conduct of the study.
* Plasma exchange 3 months prior to enrolment.
* Treatment with immunomodulatory agents others than steroids, methotrexate or azathioprine (e.g. interferon, TNF-α inhibitors) within 6 months before enrolment.
* Treatment with rituximab in the 12 months before enrolment.
* Abnormal laboratory parameters: creatinine > 1.5 times the upper normal limit (UNL), lactate dehydrogenase (LDH) > 1.5 times the UNL, C-reactive protein (CRP) > 1.5 times the UNL, hemoglobin (Hb) < 10 g/dL.
* Ongoing HIV, hepatitis C and hepatitis B infection.
* Participation in another clinical study (or use of another investigational medicinal product [IMP]) within 3 months prior to enrolment
* Not able to comply with study procedures and treatment regimen.
* Employee at the study site, or spouse/partner or relative of any study staff (e.g., investigator, sub-investigators, or study nurse).
* Pregnancy or nursing mother.
* Intention to become pregnant during the course of the study.
* Female subjects of childbearing potential either not using, or not willing to use, a medically reliable method of contraception for the entire duration of the study, or not sexually abstinent for the entire duration of the study, or not surgically sterile.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Program Director Clinical R&D, Study Director — CSL Behring
Locations (22):
- Belgium (4):
  - Study Site, Brussels
  - Study Site, Edegem
  - Study Site, Ghent
  - Study Site, Leuven
- Finland (3):
  - Study Site, Helsinki
  - Study Site, Turku
  - Study Site, Vaasa
- France (5):
  - Study Site, Limoges
  - Study Site, Lyon
  - Study Site, Marseille
  - Study Site, Montpellier
  - Study Site, Paris
- Germany (7):
  - Study Site, Berlin
  - Study Site, Feldberger Seenlandschaft
  - Study Site, Göttingen
  - Study Site, Itzehoe
  - Study Site, Prien am Chiemsee
  - Study Site, Schwedt
  - Study Site, Würzburg
- Poland (3):
  - Study Site, Krakow
  - Study Site, Lublin
  - Study Site, Wroclaw

REFERENCES:
- [Result] Leger JM, De Bleecker JL, Sommer C, Robberecht W, Saarela M, Kamienowski J, Stelmasiak Z, Mielke O, Tackenberg B, Shebl A, Bauhofer A, Zenker O, Merkies IS; PRIMA study investigators. Efficacy and safety of Privigen((R)) in patients with chronic inflammatory demyelinating polyneuropathy: results of a prospective, single-arm, open-label Phase III study (the PRIMA study). J Peripher Nerv Syst. 2013 Jun;18(2):130-40. doi: 10.1111/jns5.12017. PMID 23781960
- [Derived] Merkies ISJ, Lawo JP, Edelman JM, De Bleecker JL, Sommer C, Robberecht W, Saarela M, Kamienowski J, Stelmasiak Z, Mielke O, Tackenberg B, Leger JM; PRIMA trial investigators. Minimum clinically important difference analysis confirms the efficacy of IgPro10 in CIDP: the PRIMA trial. J Peripher Nerv Syst. 2017 Jun;22(2):149-152. doi: 10.1111/jns.12204. No abstract available. PMID 28594116

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study enrolled subjects at 13 participating study centers in 5 countries in Europe.
Pre-assignment Details: A total of 31 subjects were screened and 28 were eligible.
  * Intravenous immunoglobulin (IVIG)-untreated subjects: screening took place up to 3 weeks prior to the first IgPro10 infusion
  * IVIG-pretreated subjects: Screening took place at any time at or after the last dose of pre-study IVIG (up to 10 weeks prior to the first IgPro10 infusion)
Period: Overall Study
Arm/Group | IgPro10
Started | 28
Completed | 25
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Insufficient response | 1

BASELINE CHARACTERISTICS:
Arm/Group | IgPro10
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 18
Previous IVIG treatment [Number; unit: participants]
  IVIG-pretreated subjects | 13
  IVIG-untreated subjects | 15

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate
Description: Percentage of responders based on the adjusted Inflammatory Neuropathy Cause and Treatment Scale (INCAT) score.
  Responders were defined as those subjects who: 1) demonstrated a "clinically meaningful improvement" between baseline and Week 25, or 2) who were discontinued from the study for any reason after the start of IgPro10 treatment but with "clinically meaningful improvement" at the last study visit.
  "Clinically meaningful improvement" was a decrease of at least 1 adjusted INCAT score point excluding an improvement of one point in the total score if this improvement was only due to a decrease in the upper limb score of 1 to 0.
Time Frame: 25 weeks
Population: The full analysis set (FAS) includes all subjects who received at least one dose of IgPro10, regardless of whether or not the subject recorded an efficacy variable measurement. The valid cases set (VCS) consists of all FAS subjects without any major protocol deviation (ie, the subjects who participated in the study as intended).
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | IgPro10
Number analyzed (Participants) | 28
percentage of responders
  FAS (n = 28) | 60.7 [42.409 to 76.434]
  VCS (n = 22) | 63.6 [42.952 to 80.267]

2. Secondary Outcome: Change in Adjusted INCAT Score
Description: The change in INCAT score was determined at the completion visit compared to baseline and to the last measurement under the previous IVIG treatment using a non-parametric analysis to calculate the Hodges-Lehmann point estimate and the corresponding Tukey confidence interval on an exploratory basis.
  The INCAT disability score ranges from 0 to 10 and is the sum of arm and leg disability each rated between 0 and 5 (where arm = 0 indicates 'no upper limb problems' and arm = 5 indicates 'inability to use either arm for any purposeful movement', and leg = 0 indicates 'walking not affected', and leg = 5 indicates 'restricted to wheelchair, unable to stand and walk a few steps with help'). Thus, a higher INCAT disability score indicates greater disability. Negative values for change in INCAT score indicate improvement, with a more negative value indicating greater improvement compared with the value at baseline.
Time Frame: Up to 34 weeks
Population: The FAS includes all subjects who received at least one dose of IgPro10, regardless of whether or not the subject recorded an efficacy variable measurement. Analysed subgroups include all subjects and IVIG-pretreated and IVIG-untreated subjects from baseline to completion, and IVIG-pretreated subjects from last IVIG treatment to completion.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 28
score on a scale
  All subjects; n = 28 | -1.3 [-2.0 to -0.5]
  IVIG-pretreated; n = 13 | -2.0 [-2.5 to -1.0]
  IVIG-untreated; n = 15 | -1.0 [-2.0 to 0.0]
  IVIG-pretreated (last IVIG to completion); n = 13 | -2.0 [-2.5 to -1.0]

3. Secondary Outcome: Change in Maximum Grip Strength
Description: Change in maximum grip strength of the dominant hand. A non-parametric analysis was used to calculate the Hodges-Lehmann point estimate and the corresponding Tukey confidence interval on an exploratory basis. Positive values for change in maximum grip strength indicate improvement.
Time Frame: Up to 34 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: kPa
Arm/Group | IgPro10
Number analyzed (Participants) | 28
kPa
  All subjects; n = 28 | 9.0 [-1.0 to 22.3]
  IVIG-pretreated; n = 13 | 8.0 [-5.0 to 25.0]
  IVIG-untreated; n = 15 | 9.0 [-6.0 to 35.0]
  IVIG-pretreated (last IVIG to completion); n = 13 | -1.5 [-12.5 to 14.5]

4. Secondary Outcome: Change in Medical Research Council Sum Scale (MRC)
Description: The change in MRC sum score was determined at the completion visit compared to baseline and to the last measurement under the previous IVIG treatment using a non-parametric analysis to calculate the Hodges-Lehmann point estimate and the corresponding Tukey confidence interval on an exploratory basis.
  The 80-point MRC sum score is the sum of scores for eight bilateral (left and right side) muscle groups, each rated between 0 (no visible contraction) to 5 (normal movement). A higher MRC sum score indicates greater muscle contraction/limb movement. Positive values for change in MRC sum score indicate improvement, with a more positive value indicating greater muscle contraction/ limb movement compared with the value at baseline.
Time Frame: Up to 34 weeks
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | IgPro10
Number analyzed (Participants) | 28
score on a scale
  All subjects; n = 28 | 6.5 [4.0 to 9.5]
  IVIG-pretreated; n = 13 | 6.0 [2.5 to 10.0]
  IVIG-untreated; n = 15 | 7.0 [3.0 to 12.5]
  IVIG-pretreated (last IVIG to completion); n = 13 | 1.0 [-2.5 to 4.5]

5. Secondary Outcome: Immunoglobulin G (IgG) Level
Time Frame: At baseline and at Weeks 7, 13 and 19 (levels determined immediately before and after IVIG infusion), and at completion visit (Week 25)
Population: The FAS includes all subjects who received at least one dose of IgPro10, regardless of whether or not the subject recorded an efficacy variable measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- IgPro10 - Before Infusion: IgG levels were determined before infusion with IgPro10.
- IgPro10 - After Infusion: IgG levels were determined after infusion with IgPro10.
Arm/Group | IgPro10 - Before Infusion | IgPro10 - After Infusion
Number analyzed (Participants) | 28 | 27
mg/dL
  At baseline (n = 28 and 27, respectively) | 1259.5 (377.47) | 2859.2 (846.83)
  At Week 7 (n = 26) | 1750.0 (313.73) | 3228.8 (803.22)
  At Week 13 (n = 25) | 1733.2 (353.00) | 3496.7 (575.11)
  At Week 19 (n = 25 and 24, respectively) | 1684.6 (306.62) | 3386.1 (567.05)
  At Completion (n = 0 and 28 respectively) | NA (NA) — There was no IgPro10 infusion at the completion visit. Thus, the IgG level measured at the completion visit represents the IgG level 3 weeks after the last infusion (at week 19) or at early discontinuation. | 1943.6 (465.85)

6. Secondary Outcome: Frequency of Adverse Events (AEs)
Description: Overall rate of AEs per infusion.
Time Frame: For the duration of the study, up to 34 weeks
Population: The safety data set (SDS) comprised all subjects treated with the study drug.
Measure: Number; unit: AE rate per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro10
Number analyzed (Participants) | 28
Number analyzed (Infusions) | 259
AE rate per infusion | 0.417

7. Secondary Outcome: Severity of AEs Per Infusion
Description: The severity of each AE was to be graded by the investigator as follows:
  * Mild: Symptoms were easily tolerated and there was no interference with daily activities.
  * Moderate: Discomfort enough to cause some interference with daily activities.
  * Severe: Incapacitating with inability to work or do usual activity.
Time Frame: For the duration of the study, up to 34 weeks
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: AE rate per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro10
Number analyzed (Participants) | 28
Number analyzed (Infusions) | 259
AE rate per infusion
  Mild AE | 0.266
  Moderate AE | 0.143
  Severe AE | 0.008

8. Secondary Outcome: Severity of AEs Per Subject
Description: as for outcome 7
Time Frame: 34 weeks
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro10
Number analyzed (Participants) | 28
percentage of subjects
  Mild AE | 67.9
  Moderate AE | 46.4
  Severe AE | 7.1

9. Secondary Outcome: Relatedness of AEs Per Infusion
Description: The causal relationship of an AE to the study drug was to be assessed and assigned by the investigator.
Time Frame: For the duration of the study, up to 34 weeks
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: AE rate per infusion
Units Other Than Participants: Infusions
Arm/Group | IgPro10
Number analyzed (Participants) | 28
Number analyzed (Infusions) | 259
AE rate per infusion
  Not Related | 0.201
  Unlikely Related | 0.027
  Possibly Related | 0.081
  Probably Related | 0.042
  Related | 0.066

10. Secondary Outcome: Relatedness of AEs Per Subject
Description: The causal relationship of an AE to the study drug was to be assessed and assigned by the investigator.
Time Frame: For the duration of the study, up to 34 weeks
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: percentage of subjects
Arm/Group | IgPro10
Number analyzed (Participants) | 28
percentage of subjects
  Not Related | 60.7
  Unlikely Related | 14.3
  Possibly Related | 39.3
  Probably Related | 25.0
  Related | 25.0

11. Secondary Outcome: Mean Change in Systolic and Diastolic Blood Pressure During Infusion
Description: Systolic and diastolic blood pressure (BP) were measured before the start of IgPro10 infusion, at 30 minutes and 1 hour after the start of infusion, then every hour until the end of infusion and at 1 hour after the end of infusion. Mean changes from the pre-infusion value to each of the post-infusion values were calculated for each infusion, and the mean value and standard deviation (SD) of these individual mean changes is reported.
Time Frame: At Days 1 to 5 and at Weeks 4, 7, 10, 13, 16, 19 and 22.
Population: The SDS comprised all subjects treated with the study drug.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | IgPro10
Number analyzed (Participants) | 28
mm Hg
  Systolic BP mean value of mean change | 1.03 (7.62)
  Diastolic BP mean value of mean change | 0.99 (7.46)

12. Secondary Outcome: Mean Change in Pulse Rate During Infusion
Description: Pulse rate was measured before the start of IgPro10 infusion, at 30 minutes and 1 hour after the start of infusion, then every hour until the end of infusion and at 1 hour after the end of infusion. Mean changes from the pre-infusion value to each of the post-infusion values were calculated for each infusion, and the mean value and SD of these individual mean changes is reported.
Time Frame: At Days 1 to 5 and at Weeks 4, 7, 10, 13, 16, 19 and 22.
Population: The SDS comprised all subjects treated with the study drug
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | IgPro10
Number analyzed (Participants) | 28
beats per minute | -1.14 (3.58)

13. Secondary Outcome: Mean Change in Body Temperature During Infusion
Description: Body temperature was measured before the start of IgPro10 infusion, at 30 minutes and 1 hour after the start of infusion, then every hour until the end of infusion and at 1 hour after the end of infusion. Mean changes from the pre-infusion value to each of the post-infusion values were calculated for each infusion, and the mean value and SD of these individual mean changes is reported.
Time Frame: At Days 1 to 5 and at Weeks 4, 7, 10, 13, 16, 19 and 22.
Population: The SDS comprised all subjects treated with the study drug.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | IgPro10
Number analyzed (Participants) | 28
°C | 0.06 (0.17)

14. Secondary Outcome: Number of Subjects With Normal/Abnormal Not Clinically Significant (ANCS) Value at Baseline Changing to Abnormal Clinically Significant (ACS) Value at Completion Visit in Routine Laboratory Parameters.
Description: Number of subjects with changes from normal/ANCS values at baseline to ACS values at Completion Visit in routine laboratory parameters including hematology and serum chemistry analytes. Investigators flagged each laboratory value as normal, ANCS or ACS at each assessment timepoint.
Time Frame: At Day 1 (baseline) and at Completion Visit (Week 25 or early discontinuation)
Population: The SDS comprised all subjects treated with the study drug.
Measure: Number; unit: participants
Arm/Group | IgPro10
Number analyzed (Participants) | 28
participants | 4

ADVERSE EVENTS:
Time Frame: For the duration of the study, up to 34 weeks.
Description: Only AEs starting at or after the first study drug infusion are included. The safety data set (SDS) comprised all subjects treated with the study drug.
Arm/Group | IgPro10
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 22/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=28)
Haemolysis (Blood and lymphatic system disorders) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IgPro10 (N=28)
Leukopenia (Blood and lymphatic system disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3)
Asthenia (General disorders) | 4 (4)
Influenza-like illness (General disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Headache (Nervous system disorders) | 9 (20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.